CLINICAL TRIAL: NCT06940453
Title: Clinical/Radiological Outcomes Associated With CONDUIT™ Anterior Lumbar Interbody Fusion (ALIF) Cage System With Supplemental Fixation for Treatment of Lumbar Degenerative Disc Disease at One or Two Contiguous Spinal Levels From L2-S1
Brief Title: CONDUIT™ Anterior Lumbar Interbody Fusion (ALIF) Cage System in Lumbar Degenerative Disease
Status: Recruiting | Type: Observational
Sponsor: University College Dublin (Other)
Collaborators: Mater Misericordiae University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CONDUIT™
Record Dates: First submitted 2024-07-09; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-07

CONDITIONS: Lumbar Degenerative Disease
Keywords: INTERBODY FUSION; SPINE SURGERY; LUMBAR DEGENERATION; SPINAL FUSION; SPINAL FIXATION
MeSH Terms: interventions — Urinary Diversion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- SYNFIX COHORT: This cohort will be composed of historical, retrospective data (70 patients total) of patients who underwent surgical stabilisation for lumbar degenerative disease using the SYNFIX system, with supplemental posterior fixation.
  Interventions: Device: CONDUIT

INTERVENTIONS:
Device: CONDUIT — Arm Description: Group/Cohort Description: This cohort is composed of patients who will be prospectively enrolled (35 total). These patients will undergo spinal stabilisation for lumbar degenerative disease using the CONDUIT ALIF cage system with supplemental posterior fixation. This device is FDA approved thus this is post market observational intervention.

SUMMARY:
This will be a prospective, multi-centre study at a National Tertiary Referral Centre for spinal trauma and spinal cord injuries, serving a catchment area of 5 million people. This study will follow patients undergoing anterior lumbar interbody fusion (ALIF) procedure. This trial seeks to evaluate the performance of this CE-marked device, and to assess outcomes in frail and non-frail patient cohorts. The CONDUIT™ ALIF Cage System are intervertebral body fusion devices intended for use for anterior lumbar interbody fusion in skeletally mature patients. The devices are 3D printed cellular titanium implants that feature 80% porous macro-, micro- and nanostructures, are designed to mimic cortical and cancellous bone, and facilitate fusion. This pilot study hypothesizes that the use of CONDUIT ALIF Cage system to treat lumbar degenerative disc disease will achieve results comparable to historical cases using SYNFIX Systems.

DETAILED DESCRIPTION:
This will be a prospective, multi-centre study at a National Tertiary Referral Centre for spinal trauma and spinal cord injuries, serving a catchment area of 5 million people. This study will follow patients undergoing anterior lumbar interbody fusion (ALIF) procedure at the Mater Misericordiae University and Mater Private Hospitals using the CONDUIT™ ALIF Cage System. This trial seeks to evaluate the performance of this CE-marked device, and to assess outcomes in frail and non-frail patient cohorts. The CONDUIT™ ALIF Cage System are intervertebral body fusion devices intended for use for anterior lumbar interbody fusion in skeletally mature patients. The devices are 3D printed cellular titanium implants that feature 80% porous macro-, micro- and nanostructures, are designed to mimic cortical and cancellous bone, and facilitate fusion.

In spine fusion procedures, bone is encouraged to grow in order to fuse vertebrae of the spine together to relieve pain or increase stability. The likelihood of a successful fusion is thought to be influenced by multiple factors. Patient-related factors influencing fusion success include comorbidities such as osteoporosis or osteopenia, diabetes, and obesity. Factors affecting the inflammatory response, such as rheumatoid arthritis or long-term steroid use may also increase the likelihood of fusion failure. Fusion success can also be influenced by age, frailty, functional status, history of smoking or steroid use. The surgical approach may also affect fusion rate. It is thought that a posterior approach may result in higher fusion failure rates (20-30%. However, the posterior approach may be considered more appropriate for older patients with multilevel fusion, who may have a higher rate of comorbidities which affect fusion rate.

Frailty is a clinically recognizable syndrome comprised of declining physiological reserve, characterized by decreased resilience to adverse health outcomes. Fried et al have defined frailty as meeting three out of five of the following criteria: low grip strength, low energy, slow walking speed, low physical activity, unintentional weight loss. The modified 5-item frailty index (mFI-5) is another method of measuring frailty commonly used in clinical settings. It has been shown to predict the occurrence of adverse outcomes following various orthopaedic surgeries. The five comorbidities included in the mFI-5 are a history of hypertension, COPD, diabetes mellitus, congestive heart failure, and a non-independent functional status. This pilot study hypothesizes that the use of CONDUIT ALIF Cage system to treat lumbar degenerative disc disease will achieve results comparable to historical cases using SYNFIX Systems.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old
* Consenting patients undergoing anterior lumbar interbody fusion (ALIF) procedure whom the Conduit cage system is appropriate will be included in this study.

Exclusion Criteria:

* Patients under 18 years of age
* Non-surgical candidates, patients with contraindications to surgery (e.g. medical comorbidities, known infection, pregnancy etc.),
* Patients with established osteoporosis
* Long-term, systemic steroid use
* Systemic diseases (e.g. rheumatoid arthritis, AIDS, HIV, etc.),
* Patients unwilling or unable to give informed consent, or patients unwilling or unable to complete Health-related quality of (HRQOL) outcome life measures at the specified study time points pre- and post-operatively.
* Subjects who have a history of drug or alcohol use that, in the opinion of the investigator, would interfere with adherence to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years old) with lumbar degenerative disease requiring surgical intervention and stabilisation with instrumentation
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Radiographic Fusion at 24 months as inferred by Presence of Segmental Stability and Absence of Mechanical Failure on Xray/CT | 24 months
  The primary objective of this study is to evaluate the radiographic assessment of fusion at 24 months postoperatively. This radiographic assessment will consist of plain Xrays preoperatively, at 6 weeks, 3 months, 6 months and 24 months postoperatively. These will include a combination of anterior, lateral, flexion and extension views images of lumbar spine used to infer stability.
  Fusion failure (pseudarthrosis) will be defined as signs of mechanical failure (such as peri-implant radiolucency/haloing, screw/rod fracture, etc.) or <50% bridging trabecular bone on CT scan at 12 months postoperatively. Assessment of fusion will be conducted by a musculoskeletal radiologist and 2 independent fellowship trained spine surgeons.

SECONDARY OUTCOMES:
Changes in Patient Reported Pain as Measured Using Visual Analogue Scale Score Throughout Follow up Period | 24 months
  At predetermined intervals (preoperative, at time of discharge and 6 weeks, 3 months, 6 months, 12 months and 24 months follow up), subjective patient pain will be recorded using the Visual Analogue Scale which ranges from 0 to 10 with a score of 10 indicating the most severe possible pain and a score of 0 indicating no pain is present.
  A secondary objective of this study is to prospectively gather patient reported outcomes (PROMs) in terms of pain and function
Changes in Patient Reported Function as Measured Using Oswestry Disability Index Throughout Follow up Period | 24 months
  At predetermined intervals (preoperative, at time of discharge and 6 weeks, 3 months, 6 months, 12 months and 24 months follow up), subjective patient function will be recorded using the Oswestry Disability Index which ranges from 0 to 100 disability with a score of 100% indicating complete disability rendering a patient bed bound and a score of 0% indicating minimal disability is present.
Changes in Patient Reported Function as Measured Using Short Form 12 Throughout Follow up Period | 24 months
  At predetermined intervals (preoperative, at time of discharge and 6 weeks, 3 months, 6 months, 12 months and 24 months follow up), subjective patient function will be recorded using the Short Form 12 which returns component scores representing both physical and mental status. These scores are adjusted and compare versus averages within the United States population. Both scores have an average score of 50 with a standard deviation of 10. Lower scores indicate worse function while higher scores indicate greater function.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Butler, PhD, Principal Investigator — Mater Misericordiae University Hospital
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: No
Analysis / breakdown of IPD is not felt to benefit study results or outcomes based on the study methodology.

REFERENCES:
- [Background] Verla T, Xu DS, Davis MJ, Reece EM, Kelly M, Nunez M, Winocour SJ, Ropper AE. Failure in Cervical Spinal Fusion and Current Management Modalities. Semin Plast Surg. 2021 Feb;35(1):10-13. doi: 10.1055/s-0041-1722853. Epub 2021 May 10. PMID 33994872
- [Background] Lau D, Chou D, Ziewacz JE, Mummaneni PV. The effects of smoking on perioperative outcomes and pseudarthrosis following anterior cervical corpectomy: Clinical article. J Neurosurg Spine. 2014 Oct;21(4):547-58. doi: 10.3171/2014.6.SPINE13762. Epub 2014 Jul 11. PMID 25014499
- [Background] undefined
- [Background] Badiee RK, Mayer R, Pennicooke B, Chou D, Mummaneni PV, Tan LA. Complications following posterior cervical decompression and fusion: a review of incidence, risk factors, and prevention strategies. J Spine Surg. 2020 Mar;6(1):323-333. doi: 10.21037/jss.2019.11.01. PMID 32309669